CLINICAL TRIAL: NCT03765762
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Tolerability of Pulsed GRF6019 Infusions in Subjects With Severe Alzheimer's Disease
Brief Title: A Study to Assess the Safety of GRF6019 Infusions in Subjects With Severe Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Alkahest study 6019-202
Record Dates: First submitted 2018-11-29; First posted 2018-12-05 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2019-05

CONDITIONS: Severe Alzheimer Disease
Keywords: Brain Diseases; Nervous System Diseases; Central Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Dementia; Tauopathy
MeSH Terms: conditions — Alzheimer Disease; Brain Diseases; Nervous System Diseases; Central Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders; Dementia; Tauopathies | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GRF6019 (Experimental): Subjects will receive intravenously 250 mL of GRF6019 each day for 5 consecutive days.
  Interventions: Drug: GRF6019
- Placebo (Placebo Comparator): Subjects will receive intravenously 250 mL of placebo each day for 5 consecutive days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GRF6019 — GRF6019 for IV infusion
  Arms: GRF6019
Other: Placebo — Placebo for IV infusion
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, and potential cognitive benefit of the experimental treatment GRF6019 in subjects with severe Alzheimer's disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study to assess the safety, tolerability and potential cognitive benefit of GRF6019, a human plasma protein fraction. GRF6019 or placebo will be administered intravenously to subjects with severe Alzheimer's disease every day for 5 consecutive days. The total study duration for each subject is approximately 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD according to the National Institute on Aging-Alzheimer's Association (NIA-AA) Criteria
* MMSE Score 0-10 inclusive
* Modified Hachinski Ischemia Scale (MHIS) score of 4 or less
* Provided a signed and dated informed consent form (either the subject and/or subject's legal representative)

Exclusion Criteria:

* Evidence of clinically relevant neurological disorder(s) other than probable AD
* History of blood coagulation disorders or hypercoagulability; any concurrent use of an anticoagulant therapy. (e.g., heparin, warfarin, thrombin inhibitors, Factor Xa inhibitors). Use of antiplatelet drugs (e.g., aspirin or clopidogrel) is acceptable.
* Unstable coronary heart disease, e.g. myocardial infarction or severe or unstable angina in the 6 months prior to dosing.
* Moderate to severe congestive heart failure (New York Association Class III or IV).
* Poorly controlled high blood pressure (systolic blood pressure of 160 mmHg or higher and/or diastolic blood pressure of 100 mmHg or higher) despite treatment during the 3 months prior to dosing, or treatment refractory high blood pressure, defined as treatment requiring 3 or more antihypertensives from different classes.
* Prior hypersensitivity reaction to any human blood product or intravenous infusion; any known clinically significant drug allergy.
* Treatment with any human blood product, including transfusions and intravenous immunoglobulin, during the 6 months prior to screening.
* History of immunoglobulin A (IgA), haptoglobulin or C1 inhibitor deficiency; stroke, anaphylaxis, or thromboembolic complications of intravenous immunoglobulins.
* Hemoglobin <10 g/dL in women; and <11 g/dL in men.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Program Physician, Study Director — Alkahest, Inc.
Locations (6):
- United States (6):
  - Cognitive Clinical Trials, Gilbert, Arizona
  - Cognitive Clinical Trials, Mesa, Arizona
  - Cognitive Clinical Trials, Phoenix, Arizona
  - Pacific Research Network, San Diego, California
  - Riverside Clinical Research, Edgewater, Florida
  - Bio Behavioral Health, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- GRF6019: GRF6019 250 mL IV for 5 consecutive days
- Placebo: Placebo 250 mL IV for 5 consecutive days
Period: Overall Study
Arm/Group | GRF6019 | Placebo
Started | 18 | 8
Completed | 18 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GRF6019 | Placebo | Total
Number analyzed (Participants) | 18 | 8 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.2 (8.25) | 69.5 (8.12) | 73.5 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 7 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 8 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 8 | 26
Duration of Alzheimer's Disease [Mean (Standard Deviation); unit: years] — Years of Alzheimer's Disease Duration calculated from Medical History Year of Diagnosis to Year of Informed Consent
  years | 5.0 (1.81) | 6.0 (3.59) | 5.3 (2.46)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Treatment-emergent Adverse Events (Safety)
Description: Number of Subjects with at Least One Treatment-emergent adverse event by MedDRA preferred term and grouped by MedDRA System Organ Class
Time Frame: 5 weeks
Population: Safety: All subjects who received any amount of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6019 | Placebo
Number analyzed (Participants) | 18 | 8
Participants | 8 | 3

2. Primary Outcome: Tolerability of GRF6019
Description: Tolerability of treatment defined by the number of subjects completing 4 weeks of study after receiving 5 daily infusions
Time Frame: 5 weeks
Population: Safety: All subjects who received any amount of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6019 | Placebo
Number analyzed (Participants) | 18 | 8
Participants | 18 | 8

3. Secondary Outcome: The Mini-Mental State Examination (MMSE) Score
Description: Mean change from Baseline to 5 Weeks in the Mini-Mental State Examination (MMSE) score. The MMSE consists of 5 components: orientation to time and place, registration of 3 words, attention and calculation, recall of 3 words, and language. The scores from the 5 components are summed to obtain the overall MMSE total score. The MMSE total score can range from 0 to 30, with higher scores indicating better mental status.
Time Frame: Baseline and 5 weeks
Population: Evaluable: Subjects who received at least 4 of the 5 planned infusions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 | Placebo
Number analyzed (Participants) | 18 | 8
score on a scale | 1.3 (3.53) | 1.8 (3.20)

4. Secondary Outcome: Severe Impairment Battery (SIB) Total Score
Description: Mean change from baseline in the SIB total score. The SIB assesses cognition; test questions measure orientation, attention, language, praxis, visuospatial perception, construction, memory, orientation to name, and social interaction. There are 57 items and the range of possible scores is 0-133. Lower scores indicate greater cognitive impairment.
Time Frame: Baseline and 5 weeks
Population: Evaluable: Subjects who received at least 4 of the 5 planned infusions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 | Placebo
Number analyzed (Participants) | 18 | 8
score on a scale | 6.7 (7.59) | 10.4 (4.93)

5. Secondary Outcome: Alzheimer's Disease Cooperative Study Group Activities of Daily Living Inventory for Severe Alzheimer's Disease (ADCS-ADL-Severe)
Description: Mean change from baseline in the ADCS-ADL-Severe score. The ADCS-ADL-Severe contains 19 items covering physical and mental functioning and independence in self-care and assesses the competence in performing basic activities of daily living. The scores range from 0 to 54, with higher scores indicating less functional impairment.
Time Frame: Baseline and 5 weeks
Population: Evaluable: Subjects who received at least 4 of the 5 planned infusions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 | Placebo
Number analyzed (Participants) | 18 | 8
score on a scale | 1.6 (5.05) | 0.5 (4.93)

6. Secondary Outcome: Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change Plus Caregiver Input (ADCS-CGIC)
Description: Mean ADCS-CGIC score. A CGIC score is based on clinicians' observations of change in the subject's cognitive, functional, and behavioral performance since the beginning of a trial. The ADCS-CGIC is a rating of change and not of severity. It provides a semi structured format to enable clinicians to gather necessary clinical information from both the subject and informant to make a global impression of change. After completing the interviews, the clinician records the clinical impression of change on a 7-point Likert-type scale (from marked improvement to marked worsening). A score of 4 indicates no change, while scores > 4 indicate worsening and scores < 4 indicate improvement.
Time Frame: Baseline and 5 weeks
Population: Evaluable: Subjects who received at least 4 of the 5 planned infusions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 | Placebo
Number analyzed (Participants) | 18 | 8
score on a scale | 3.9 (0.83) | 4.0 (0.76)

7. Secondary Outcome: Neuropsychiatric Inventory Nursing Home (NPI-NH) Total Score
Description: Mean change from Baseline to 5 weeks in the NPI-NH total score. The NPI-NH is a questionnaire that quantifies behavioral changes in dementia in nursing home patients and evaluates 12 behavioral domains (Delusions, Hallucinations, Agitation/Aggression, Depression/Dysphoria, Anxiety, Elation/Euphoria, Apathy/Indifference, Disinhibition, Irritability/Lability, Aberrant Motor Behavior, Sleep and Nighttime Behavior Disorders, Appetite/Eating Changes). For each of the 12 behavioral domains the Frequency (scale:1=occasionally to 4=very frequently) is multiplied by the Severity (scale:1=Mild to 3=Severe) to obtain a domain score (frequency x severity), with a possible summed total score of 0 to 144. Lower scores correspond to less severity. A negative change score from baseline indicates improvement.
Time Frame: Baseline and 5 weeks
Population: Evaluable: Subjects who received at least 4 of the 5 planned infusions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 | Placebo
Number analyzed (Participants) | 18 | 8
score on a scale | -7.0 (19.16) | -20.0 (5.66)

8. Secondary Outcome: Neuropsychiatric Inventory (NPI) Caregiver Total Score
Description: Mean change from Baseline to 5 Weeks in NPI Total Score. NPI is based on responses from the informed caregiver during an interview. It consists of 12 sub-domains (Delusions, Hallucinations, Agitation/Aggression, Dysphoria/Depression, Anxiety, Euphoria/Elation, Apathy/Indifference, Disinhibition, Irritability/Lability, Aberrant Motor, Nighttime Behavior, Appetite/Eating). For each of the 12 behavioral domains the Distress (scale:0=Not distressing at all to 5=Extreme) is multiplied by the Severity (scale:1=Mild to 3=Severe) to obtain a domain score (distress x severity), with a possible summed total score of 0 to 180. Lower scores correspond to less severity. A negative change score from baseline indicates improvement.
Time Frame: Baseline and 5 weeks
Population: Evaluable: Subjects who received at least 4 of the 5 planned infusions
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 | Placebo
Number analyzed (Participants) | 18 | 8
score on a scale | -3.7 (11.60) | 1.5 (4.32)

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | GRF6019 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/8
Other Adverse Events (participants affected / at risk) | 8/18 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRF6019 (N=18) | Placebo (N=8)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (3) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (2) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Blood creatinine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement contains language that restricts the PI from discussing or publishing Sponsor confidential and/or proprietary information. The embargo period may be extended by mutual agreement of the Sponsor and PI.

DOCUMENTS (2):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT03765762/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03765762/SAP_001.pdf